CLINICAL TRIAL: NCT00845624
Title: DURATION OF TIME OUTSIDE, BELOW, AND ABOVE THE TARGETED Oxygen SATURATION RANGE In Preterm Infants
Brief Title: Time Outside Target Oxygen Saturation Range in Preterm Infants and Long Term Outcomes and Preterm Infants
Acronym: SAT01ROP
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, David A Kaufman, MD, University of Virginia
Other Study IDs: 12213
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2009-02

CONDITIONS: Retinopathy of Prematurity
Keywords: oxygen saturation; retinopathy of prematurity; long term outcomes; hypoxia; hyperoxia
MeSH Terms: conditions — Retinopathy of Prematurity; Hypoxia; Hyperoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Preterm infants <1500 grams or 32 weeks gestation.

SUMMARY:
The purpose of this study is to determine if there is a relationship between time spent out the targeted oxygen saturation range in preterm infants is associated with long-term outcomes such as Retinopathy of Prematurity.

DETAILED DESCRIPTION:
All infants who had a birth weight of less than 1500 grams or less than 32 weeks gestation admitted to our neonatal intensive care unit (NICU) were eligible for the study. All infants were placed on Nellcor N600 pulsoximetry. Saturation data in two-second sampling from N600 OXIMAX pulse oximeters (Covidian, CA) was collected using a modified Nellcor® Oxinet® III system (Covidian, CA and Cardiopulmonary, Milford, CT) Alarm limits were set at 83% and 93% while infants required oxygen supplementation and 85% to 100% when neonates were in room air. Desaturation events were defined as number of times the saturation fell below the low saturation limit set on the monitor (83% if oxygen requirement >21%, 85% if patient on room air). High saturation events were defined as the number of times the patient's saturation was above the upper saturation limit (93% if oxygen requirement >21%)

The data collection system summarized each day in tabular form including average SPO2, number of low and high SPO2 events, duration of events in minutes, and the percentage of time infants spent outside of the intended saturation range. Primary outcome was threshold ROP requiring laser ablation. Data on ROP was collected during hospitalization and after discharge until resolution of ROP by pediatric ophthalmologist blinded to the study results. Secondary outcomes included bronchopulmonary dysplasia, length of hospitalization, sepsis, focal bowel perforation, necrotizing enterocolitis (stage 2 or greater), patent ductus ligation, intracranial hemorrhage, and number of red blood cell and platelet transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants <1500 grams or <32 weeks gestation

Exclusion Criteria:

* None

Ages: 1 Day to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: NICU patients at risk for ROP
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Retinopathy of prematurity | 4 weeks to 52 weeks of life

SECONDARY OUTCOMES:
Time outside targeted saturation range | entire hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: David Kaufman, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Neonatal Intensive Care Unit, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Kaufman DA, Cuff AL, Wamstad JB, Boyle R, Gurka MJ, Grossman LB, Patrick P. Fluconazole prophylaxis in extremely low birth weight infants and neurodevelopmental outcomes and quality of life at 8 to 10 years of age. J Pediatr. 2011 May;158(5):759-765.e1. doi: 10.1016/j.jpeds.2010.11.002. Epub 2010 Dec 18. PMID 21168853